CLINICAL TRIAL: NCT00671918
Title: A Phase 3, Prospective, Open-Label, Multicenter Comparison Study of Lymphoseek® and Vital Blue Dye as Lymphoid Tissue Targeting Agents in Patients With Known Melanoma or Breast Cancer Who Are Undergoing Lymph Node Mapping
Brief Title: Trial of Lymphoseek in Intraoperative Localization of Lymph Nodes in Breast Cancer and Melanoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Navidea Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEO3-05
Record Dates: First submitted 2008-04-30; First posted 2008-05-05 (Estimated); Results first posted 2013-06-03 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Breast Cancer; Melanoma
Keywords: breast cancer; lymph nodes; melanoma; surgery
MeSH Terms: conditions — Breast Neoplasms; Melanoma | interventions — technetium-diethylenetriaminepentaacetic acid-mannosyl-dextran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lymphoseek, Lymphatic mapping, Injection (Experimental)
  Interventions: Drug: Lymphoseek

INTERVENTIONS:
Drug: Lymphoseek — Breast Cancer: Intradermal admin of Lymphoseek: Inject 0.2-0.4 mL in multiple divided injections or a single injection overlying the intact primary tumor or excision biopsy site OR periareolar administration of Lymphoseek: Inject 0.2-.04 mL in multiple divided doses at the margin of the areola OR subareolar administration of Lymphoseek: Inject 0.2-0.4 in multiple divided injections or a single injection in subareolar area as a subcutaneous injection OR peritumor administration of Lymphoseek: Inject 2.0-4.0 mL in multiple divided injections, intraparenchemally surrounding the tumor or biopsy cavity. For melanoma pts intradermal administration of Lymphoseek: Inject 0.2-0.4 mL in multiple divided injections or a single injection overlying the intact primary tumor or excision biopsy site.
  Other Names: technetium Tc 99m tilmanocept

SUMMARY:
Data from this pivotal clinical trial will be used to support a marketing application (i.e., NDA) for Navidea's Lymphoseek for use in intraoperative localization of lymph tissue (nodes) in the lymphatic pathway draining the primary site of a tumor.

DETAILED DESCRIPTION:
In patients with primary melanoma and breast cancer, lymph node status is often a strong predictor of outcome and influences the course of treatment a patient may follow after surgery. In an effort to reduce the morbidity and costs of detection of lymph node metastases, surgical oncologists have developed a method by which the sentinel lymph node (the first node in a draining basin) is identified intraoperatively and removed. This technique, called sentinel node biopsy, has extremely high negative predictive values for melanoma metastases and breast cancer metastases. The two largest trials for melanoma, Morton, et al (2005) and Rossi, et al (2006), reported false negative rates of 6.3% and 14.7%, respectively. Morton, et al (2006), in perhaps the most mature trial reported to date, showed a false negative rate of 3.4% . There is growing evidence that sentinel node biopsy will have a significant impact on the management of melanoma. Sentinel node biopsy also has extremely high negative predictive values for breast cancer metastases; the false-negative rates range from 0% to 9%. There is growing evidence that sentinel node biopsy will have a significant impact on the management of breast cancer. Although the survival and local recurrence studies have yet to be completed, the technique has emerged into common practice.

Lymphatic mapping with a radiopharmaceutical is a nuclear medicine examination which identifies for the surgeon the first lymph node to receive lymphatic flow from the primary tumor site. This node is removed and analyzed for the presence of malignant cells. By locating the lymph node prior to surgery, a small incision can be used to remove the node and a smaller dissection can be employed. The high negative predictive value of the technique seems to provide an accurate staging procedure and may spare patients who are lymph node negative the morbidity of a complete lymph node dissection. Consequently, staging of melanoma by lymph node mapping and biopsy may be equivalent to regional node dissection without the attendant post surgical morbidity.

An ideal lymph node imaging agent would exhibit rapid clearance from the injection site, rapid uptake and high retention within the first draining lymph node, and low uptake by the remaining lymph nodes. The ideal agent would also have low radiation absorption; high biological safety; convenient, rapid, and stable technetium-99m labeling; and biochemical purity.

Lymphoseek (technetium-99m-labeled diethylenetriamine pentaacetic acid-mannosyl-dextran, [Tc-99m]DTPA-mannosyl-dextran) is a radiotracer that accumulates in lymphatic tissue by binding to a mannose-binding protein that resides on the surface of dendritic cells and macrophages. Lymphoseek is a macromolecule consisting of multiple units of DTPA and mannose, each synthetically attached to a 10 kilodalton dextran backbone. The mannose acts as a substrate for the receptor, and the DTPA serves as a chelating agent for labeling with Tc-99m.

ELIGIBILITY:
Inclusion Criteria:

* The patient has provided written informed consent with HIPAA authorization before participating in the study, as has his/her responsible caregiver, if applicable.
* The patient is a candidate for surgical intervention, with lymph node mapping being a part of the surgical plan.
* The patient is at least 18 years of age at the time of consent.
* The patient has an ECOG performance status of Grade 0 - 2 [8].
* The patient has a clinical negative node status at the time of study entry.
* If of child bearing potential, the patient has a negative pregnancy test within 72 hours prior to administration of Lymphoseek, has been surgically sterilized, or has been postmenopausal for at least 1 year.
* The patient is currently not participating in another investigational drug study.

Melanoma Patients

* The patient has a diagnosis of primary melanoma.

Breast Cancer Patients

* The patient has a diagnosis of primary breast cancer.
* Patients with pure ductal carcinoma in situ (DCIS) or non-invasive carcinoma if lymph node biopsy is part of the surgical plan.

Exclusion Criteria:

* The patient is pregnant or lactating;
* The patient has clinical or radiological evidence of metastatic cancer including palpably abnormal or enlarged lymph nodes (i.e., all patients should be any T,N0,M0);
* The patient has a known hypersensitivity to Lymphazurin or Patent Bleu V.

Melanoma Patients

* The patient has a tumor with a Breslow depth less than 0.75mm.;
* Patients that have had preoperative chemotherapy, immunotherapy or radiation therapy;
* Patients diagnosed with a prior invasive melanoma that would occur on the same body region or potentially draining to the same nodal basin or patients with truncal or extremity primary melanoma who has had a prior breast cancer potentially draining to the same axillary nodal basin;
* Patients who have undergone node basin surgery of any type or radiation to the nodal basin(s) potentially draining the primary melanoma;
* Patients who have undergone a wide excision for their primary melanoma (>1 cm in dimension) or complex reconstruction (rotation, free flap or skin graft of any type).

Breast Cancer Patients

* The patient has bilateral primary breast cancers or multiple tumors within their breast;
* Patients that have had prior surgical procedures such as breast implants, reduction mammoplasty or axillary surgery;
* Patients scheduled for bilateral mastectomy for any reason;
* Patients that have had preoperative radiation therapy to the affected breast or axilla

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2008-04; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Orahood, M.D., Study Director — Navidea Biopharmaceuticals
Locations (15):
- United States (14):
  - Barbara Michna, M.D, Alexander City, Alabama
  - Helen Krontiras, M.D., Birmingham, Alabama
  - Anne Wallace, M.D., La Jolla, California
  - Ken Deck, M.D., Laguna Hills, California
  - Steve Martinez, M.D., Sacramento, California
  - Mark Faries, M.D., Santa Monica, California
  - Eli Avisar, M.D., Miami, Florida
  - Charles Cox, M.D., Tampa, Florida
  - Vernon Sondak, M.D., Tampa, Florida
  - Julian Kim, M.D., Cleveland, Ohio
  - Bruce Averbook, M.D, Cleveland, Ohio
  - Stephen Povoski, M.D., Columbus, Ohio
  - Thomas Frazier, M.D., Bryn Mawr, Pennsylvania
  - Ned Carp, M.D., Philadelphia, Pennsylvania
- Schlomo Schneebaum, M.D., Tel Aviv, Israel

REFERENCES:
- [Background] Morton DL, Thompson JF, Cochran AJ, Mozzillo N, Elashoff R, Essner R, Nieweg OE, Roses DF, Hoekstra HJ, Karakousis CP, Reintgen DS, Coventry BJ, Glass EC, Wang HJ; MSLT Group. Sentinel-node biopsy or nodal observation in melanoma. N Engl J Med. 2006 Sep 28;355(13):1307-17. doi: 10.1056/NEJMoa060992. PMID 17005948
- [Background] Giuliano AE, Kirgan DM, Guenther JM, Morton DL. Lymphatic mapping and sentinel lymphadenectomy for breast cancer. Ann Surg. 1994 Sep;220(3):391-8; discussion 398-401. doi: 10.1097/00000658-199409000-00015. PMID 8092905
- [Background] Morton DL, Cochran AJ, Thompson JF, Elashoff R, Essner R, Glass EC, Mozzillo N, Nieweg OE, Roses DF, Hoekstra HJ, Karakousis CP, Reintgen DS, Coventry BJ, Wang HJ; Multicenter Selective Lymphadenectomy Trial Group. Sentinel node biopsy for early-stage melanoma: accuracy and morbidity in MSLT-I, an international multicenter trial. Ann Surg. 2005 Sep;242(3):302-11; discussion 311-3. doi: 10.1097/01.sla.0000181092.50141.fa. PMID 16135917
- [Background] Rossi CR, De Salvo GL, Trifiro G, Mocellin S, Landi G, Macripo G, Carcoforo P, Ricotti G, Giudice G, Picciotto F, Donner D, Di Filippo F, Montesco MC, Casara D, Schiavon M, Foletto M, Baldini F, Testori A. The impact of lymphoscintigraphy technique on the outcome of sentinel node biopsy in 1,313 patients with cutaneous melanoma: an Italian Multicentric Study (SOLISM-IMI). J Nucl Med. 2006 Feb;47(2):234-41. PMID 16455628
- [Background] Albertini JJ, Lyman GH, Cox C, Yeatman T, Balducci L, Ku N, Shivers S, Berman C, Wells K, Rapaport D, Shons A, Horton J, Greenberg H, Nicosia S, Clark R, Cantor A, Reintgen DS. Lymphatic mapping and sentinel node biopsy in the patient with breast cancer. JAMA. 1996 Dec 11;276(22):1818-22. PMID 8946902
- [Background] Veronesi U, Paganelli G, Galimberti V, Viale G, Zurrida S, Bedoni M, Costa A, de Cicco C, Geraghty JG, Luini A, Sacchini V, Veronesi P. Sentinel-node biopsy to avoid axillary dissection in breast cancer with clinically negative lymph-nodes. Lancet. 1997 Jun 28;349(9069):1864-7. doi: 10.1016/S0140-6736(97)01004-0. PMID 9217757
- [Background] Giuliano AE, Jones RC, Brennan M, Statman R. Sentinel lymphadenectomy in breast cancer. J Clin Oncol. 1997 Jun;15(6):2345-50. doi: 10.1200/JCO.1997.15.6.2345. PMID 9196149
- [Background] Krag D, Weaver D, Ashikaga T, Moffat F, Klimberg VS, Shriver C, Feldman S, Kusminsky R, Gadd M, Kuhn J, Harlow S, Beitsch P. The sentinel node in breast cancer--a multicenter validation study. N Engl J Med. 1998 Oct 1;339(14):941-6. doi: 10.1056/NEJM199810013391401. PMID 9753708
- [Background] Krag DN, Weaver DL, Alex JC, Fairbank JT. Surgical resection and radiolocalization of the sentinel lymph node in breast cancer using a gamma probe. Surg Oncol. 1993 Dec;2(6):335-9; discussion 340. doi: 10.1016/0960-7404(93)90064-6. PMID 8130940
- [Background] Krag DN. Gamma-probe-guided resection of axillary sentinel nodes. Presented at the 48th annual symposium of the Society of Surgical Oncology, March 23-25, 1995, Boston MA.
- [Background] Guiliano AE. Axillary node mapping for breast cancer. Presented at the 48th annual symposium of the Society of Surgical Oncology, March 23-25, 1995, Boston MA.
- [Background] Wallace AM, Hoh CK, Vera DR, Darrah DD, Schulteis G. Lymphoseek: a molecular radiopharmaceutical for sentinel node detection. Ann Surg Oncol. 2003 Jun;10(5):531-8. doi: 10.1245/aso.2003.07.012. PMID 12794019
- [Background] Ellner SJ, Hoh CK, Vera DR, Darrah DD, Schulteis G, Wallace AM. Dose-dependent biodistribution of [(99m)Tc]DTPA-mannosyl-dextran for breast cancer sentinel lymph node mapping. Nucl Med Biol. 2003 Nov;30(8):805-10. doi: 10.1016/j.nucmedbio.2003.10.001. PMID 14698783
- [Background] Posther KE, McCall LM, Blumencranz PW, Burak WE Jr, Beitsch PD, Hansen NM, Morrow M, Wilke LG, Herndon JE 2nd, Hunt KK, Giuliano AE. Sentinel node skills verification and surgeon performance: data from a multicenter clinical trial for early-stage breast cancer. Ann Surg. 2005 Oct;242(4):593-9; discussion 599-602. doi: 10.1097/01.sla.0000184210.68646.77. PMID 16192820
- [Background] Barnwell JM, Arredondo MA, Kollmorgen D, Gibbs JF, Lamonica D, Carson W, Zhang P, Winston J, Edge SB. Sentinel node biopsy in breast cancer. Ann Surg Oncol. 1998 Mar;5(2):126-30. doi: 10.1007/BF02303845. PMID 9527265
- [Background] O'Hea BJ, Hill AD, El-Shirbiny AM, Yeh SD, Rosen PP, Coit DG, Borgen PI, Cody HS 3rd. Sentinel lymph node biopsy in breast cancer: initial experience at Memorial Sloan-Kettering Cancer Center. J Am Coll Surg. 1998 Apr;186(4):423-7. doi: 10.1016/s1072-7515(98)00060-x. PMID 9544956
- [Background] Klimberg VS, Rubio IT, Henry R, Cowan C, Colvert M, Korourian S. Subareolar versus peritumoral injection for location of the sentinel lymph node. Ann Surg. 1999 Jun;229(6):860-4; discussion 864-5. doi: 10.1097/00000658-199906000-00013. PMID 10363900
- [Background] Borgstein PJ, Meijer S, Pijpers RJ, van Diest PJ. Functional lymphatic anatomy for sentinel node biopsy in breast cancer: echoes from the past and the periareolar blue method. Ann Surg. 2000 Jul;232(1):81-9. doi: 10.1097/00000658-200007000-00012. PMID 10862199
- [Background] Smith LF, Cross MJ, Klimberg VS. Subareolar injection is a better technique for sentinel lymph node biopsy. Am J Surg. 2000 Dec;180(6):434-7; discussion 437-8. doi: 10.1016/s0002-9610(00)00521-3. PMID 11182393
- [Background] Tsugawa K, Noguchi M, Miwa K, Bando E, Yokoyama K, Nakajima K, Michigishi T, Tonami N, Minato H, Nonomura A. Dye- and gamma probe-guided sentinel lymph node biopsy in breast cancer patients: using patent blue dye and technetium-99m-labeled human serum albumin. Breast Cancer. 2000 Jan;7(1):87-94. doi: 10.1007/BF02967195. PMID 11029778
- [Background] Donahue EJ. Sentinel node imaging and biopsy in breast cancer patients. Am J Surg. 2001 Oct;182(4):426-8. doi: 10.1016/s0002-9610(01)00731-0. PMID 11720685
- [Background] Martin RC, Derossis AM, Fey J, Yeung H, Yeh SD, Akhurst T, Heerdt AS, Petrek J, VanZee KJ, Montgomery LL, Borgen PI, Cody HS 3rd. Intradermal isotope injection is superior to intramammary in sentinel node biopsy for breast cancer. Surgery. 2001 Sep;130(3):432-8. doi: 10.1067/msy.2001.116412. PMID 11562666
- [Background] Bauer TW, Spitz FR, Callans LS, Alavi A, Mick R, Weinstein SP, Bedrosian I, Fraker DL, Bauer TL, Czerniecki BJ. Subareolar and peritumoral injection identify similar sentinel nodes for breast cancer. Ann Surg Oncol. 2002 Mar;9(2):169-76. doi: 10.1007/BF02557370. PMID 11888875
- [Background] Kern KA. Concordance and validation study of sentinel lymph node biopsy for breast cancer using subareolar injection of blue dye and technetium 99m sulfur colloid. J Am Coll Surg. 2002 Oct;195(4):467-75. doi: 10.1016/s1072-7515(02)01312-1. PMID 12375751
- [Background] Tuttle TM, Colbert M, Christensen R, Ose KJ, Jones T, Wetherille R, Friedman J, Swenson K, McMasters KM. Subareolar injection of 99mTc facilitates sentinel lymph node identification. Ann Surg Oncol. 2002 Jan-Feb;9(1):77-81. doi: 10.1245/aso.2002.9.1.77. PMID 11829434
- [Background] Zavagno G, Meggiolaro F, Rossi CR, Casara D, Pescarini L, Marchet A, Denetto V, Baratella P, Lise M. Subareolar injection for sentinel lymph node location in breast cancer. Eur J Surg Oncol. 2002 Nov;28(7):701-4. doi: 10.1053/ejso.2002.1340. PMID 12431465
- [Background] Pelosi E, Bello M, Giors M, Ala A, Giani R, Bussone R, Bisi G. Sentinel lymph node detection in patients with early-stage breast cancer: comparison of periareolar and subdermal/peritumoral injection techniques. J Nucl Med. 2004 Feb;45(2):220-5. PMID 14960639
- [Background] Wada N, Imoto S, Yamauchi C, Hasebe T, Ochiai A, Ebihara S. Correlation between concordance of tracers, order of harvest, and presence of metastases in sentinel lymph nodes with breast cancer. Ann Surg Oncol. 2005 Jun;12(6):497-503. doi: 10.1245/ASO.2005.07.013. Epub 2005 Apr 19. PMID 15864480
- [Background] Rodier JF, Velten M, Wilt M, Martel P, Ferron G, Vaini-Elies V, Mignotte H, Bremond A, Classe JM, Dravet F, Routiot T, de Lara CT, Avril A, Lorimier G, Fondrinier E, Houvenaeghel G, Avigdor S. Prospective multicentric randomized study comparing periareolar and peritumoral injection of radiotracer and blue dye for the detection of sentinel lymph node in breast sparing procedures: FRANSENODE trial. J Clin Oncol. 2007 Aug 20;25(24):3664-9. doi: 10.1200/JCO.2006.08.4228. Epub 2007 May 7. PMID 17485709
- [Background] Hodgson N, Zabel P, Mattar AG, Engel CJ, Girvan D, Holliday R. A new radiocolloid for sentinel node detection in breast cancer. Ann Surg Oncol. 2001 Mar;8(2):133-7. doi: 10.1007/s10434-001-0133-2. PMID 11258777
- [Background] Simon R. Optimal two-stage designs for phase II clinical trials. Control Clin Trials. 1989 Mar;10(1):1-10. doi: 10.1016/0197-2456(89)90015-9. PMID 2702835
- [Background] Cox CE, Pendas S, Cox JM, Joseph E, Shons AR, Yeatman T, Ku NN, Lyman GH, Berman C, Haddad F, Reintgen DS. Guidelines for sentinel node biopsy and lymphatic mapping of patients with breast cancer. Ann Surg. 1998 May;227(5):645-51; discussion 651-3. doi: 10.1097/00000658-199805000-00005. PMID 9605656
- [Background] McMasters KM, Wong SL, Chao C, Woo C, Tuttle TM, Noyes RD, Carlson DJ, Laidley AL, McGlothin TQ, Ley PB, Brown CM, Glaser RL, Pennington RE, Turk PS, Simpson D, Edwards MJ; University of Louisville Breast Cancer Study Group. Defining the optimal surgeon experience for breast cancer sentinel lymph node biopsy: a model for implementation of new surgical techniques. Ann Surg. 2001 Sep;234(3):292-9; discussion 299-300. doi: 10.1097/00000658-200109000-00003. PMID 11524582
- [Background] Miltenburg DM, Miller C, Karamlou TB, Brunicardi FC. Meta-analysis of sentinel lymph node biopsy in breast cancer. J Surg Res. 1999 Jun 15;84(2):138-42. doi: 10.1006/jsre.1999.5629. PMID 10357910
- [Background] Kim T, Giuliano AE, Lyman GH. Lymphatic mapping and sentinel lymph node biopsy in early-stage breast carcinoma: a metaanalysis. Cancer. 2006 Jan 1;106(1):4-16. doi: 10.1002/cncr.21568. PMID 16329134
- [Background] Bergkvist L, Frisell J, Liljegren G, Celebioglu F, Damm S, Thorn M. Multicentre study of detection and false-negative rates in sentinel node biopsy for breast cancer. Br J Surg. 2001 Dec;88(12):1644-8. doi: 10.1046/j.0007-1323.2001.01948.x. PMID 11736980
- [Background] Krag DN, Meijer SJ, Weaver DL, Loggie BW, Harlow SP, Tanabe KK, Laughlin EH, Alex JC. Minimal-access surgery for staging of malignant melanoma. Arch Surg. 1995 Jun;130(6):654-8; discussion 659-60. doi: 10.1001/archsurg.1995.01430060092018. PMID 7539252
- [Background] Albertini JJ, Cruse CW, Rapaport D, Wells K, Ross M, DeConti R, Berman CG, Jared K, Messina J, Lyman G, Glass F, Fenske N, Reintgen DS. Intraoperative radio-lympho-scintigraphy improves sentinel lymph node identification for patients with melanoma. Ann Surg. 1996 Feb;223(2):217-24. doi: 10.1097/00000658-199602000-00016. PMID 8597518
- [Background] Habib FA, Lodish ME, Mittal VK, Young SC. Sentinel lymph node dissection for primary cutaneous melanoma: a community hospital's initial experience. Am Surg. 2000 Mar;66(3):291-5. PMID 10759202
- [Background] Estourgie SH, Nieweg OE, Valdes Olmos RA, Hoefnagel CA, Kroon BB. Review and evaluation of sentinel node procedures in 250 melanoma patients with a median follow-up of 6 years. Ann Surg Oncol. 2003 Jul;10(6):681-8. doi: 10.1245/aso.2003.01.023. PMID 12839854
- [Background] Vuylsteke RJ, van Leeuwen PA, Statius Muller MG, Gietema HA, Kragt DR, Meijer S. Clinical outcome of stage I/II melanoma patients after selective sentinel lymph node dissection: long-term follow-up results. J Clin Oncol. 2003 Mar 15;21(6):1057-65. doi: 10.1200/JCO.2003.07.170. PMID 12637471
- [Background] Yee VS, Thompson JF, McKinnon JG, Scolyer RA, Li LX, McCarthy WH, O'Brien CJ, Quinn MJ, Saw RP, Shannon KF, Stretch JR, Uren RF. Outcome in 846 cutaneous melanoma patients from a single center after a negative sentinel node biopsy. Ann Surg Oncol. 2005 Jun;12(6):429-39. doi: 10.1245/ASO.2005.03.074. Epub 2005 Apr 28. PMID 15886905
- [Background] Morton DL, Wen DR, Wong JH, Economou JS, Cagle LA, Storm FK, Foshag LJ, Cochran AJ. Technical details of intraoperative lymphatic mapping for early stage melanoma. Arch Surg. 1992 Apr;127(4):392-9. doi: 10.1001/archsurg.1992.01420040034005. PMID 1558490
- [Background] Reintgen D, Cruse CW, Wells K, Berman C, Fenske N, Glass F, Schroer K, Heller R, Ross M, Lyman G, et al. The orderly progression of melanoma nodal metastases. Ann Surg. 1994 Dec;220(6):759-67. doi: 10.1097/00000658-199412000-00009. PMID 7986143
- [Background] Thompson JF, McCarthy WH, Bosch CM, O'Brien CJ, Quinn MJ, Paramaesvaran S, Crotty K, McCarthy SW, Uren RF, Howman-Giles R. Sentinel lymph node status as an indicator of the presence of metastatic melanoma in regional lymph nodes. Melanoma Res. 1995 Aug;5(4):255-60. doi: 10.1097/00008390-199508000-00008. PMID 7496161
- [Background] Morton DL, Wen DR, Foshag LJ, Essner R, Cochran A. Intraoperative lymphatic mapping and selective cervical lymphadenectomy for early-stage melanomas of the head and neck. J Clin Oncol. 1993 Sep;11(9):1751-6. doi: 10.1200/JCO.1993.11.9.1751. PMID 8355042
- [Background] Karakousis CP, Velez AF, Spellman JE Jr, Scarozza J. The technique of sentinel node biopsy. Eur J Surg Oncol. 1996 Jun;22(3):271-5. doi: 10.1016/s0748-7983(96)80017-5. PMID 8654611
- [Background] Lingam MK, Mackie RM, McKay AJ. Intraoperative identification of sentinel lymph node in patients with malignant melanoma. Br J Cancer. 1997;75(10):1505-8. doi: 10.1038/bjc.1997.257. PMID 9166945
- [Result] Sondak VK, King DW, Zager JS, Schneebaum S, Kim J, Leong SP, Faries MB, Averbook BJ, Martinez SR, Puleo CA, Messina JL, Christman L, Wallace AM. Combined analysis of phase III trials evaluating [(9)(9)mTc]tilmanocept and vital blue dye for identification of sentinel lymph nodes in clinically node-negative cutaneous melanoma. Ann Surg Oncol. 2013 Feb;20(2):680-8. doi: 10.1245/s10434-012-2612-z. Epub 2012 Oct 3. PMID 23054107
- [Result] Wallace AM, Han LK, Povoski SP, Deck K, Schneebaum S, Hall NC, Hoh CK, Limmer KK, Krontiras H, Frazier TG, Cox C, Avisar E, Faries M, King DW, Christman L, Vera DR. Comparative evaluation of [(99m)tc]tilmanocept for sentinel lymph node mapping in breast cancer patients: results of two phase 3 trials. Ann Surg Oncol. 2013 Aug;20(8):2590-9. doi: 10.1245/s10434-013-2887-8. Epub 2013 Mar 17. PMID 23504141

RESULTS

PARTICIPANT FLOW:
Groups:
- Lymphoseek, Lymphatic Mapping, Injection: Melanoma and breast cancer patients to receive a single dose of 50 μg Lymphoseek radiolabeled with 0.5 or 1.0 mCi Tc-99m and blue dye for lymphatic mapping and surgical resection of lymph nodes.
Period: Overall Study
Arm/Group | Lymphoseek, Lymphatic Mapping, Injection
Started | 186
Completed | 169
Not Completed | 17

BASELINE CHARACTERISTICS:
Population: Of the 186 participants who enrolled in the trial, 179 were administered the study agent, Lymphoseek, and therefore this participant number is used for the baseline analysis.
Groups:
- Lymphoseek: Enrolled patients who were administered any injection of Lymphoseek.
Arm/Group | Lymphoseek
Number analyzed (Participants) | 179
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 120
  >=65 years | 59
Age Continuous [Mean (Standard Deviation); unit: years] | 58.5 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128
  Male | 51
Region of Enrollment [Number; unit: participants]
  United States | 161
  Israel | 18

OUTCOME MEASURES:

1. Primary Outcome: Concordance of Blue Dye and Lymphoseek
Description: The proportion of lymph nodes detected intraoperatively by blue dye that were also detected by Lymphoseek.
Time Frame: Surgery after injections of Lymphoseek and blue dye
Population: All enrolled patients who were injected with both Lymphoseek and blue dye, who underwent surgery and had at least one lymph node stained intraoperatively by blue dye, and for whom the tissue type (lymphatic/nonlymphatic) and pathology status (presence/absence of tumor cells) was confirmed.
Measure: Number (95% Confidence Interval); unit: Proportion of Lymph Nodes
Units Other Than Participants: Lymph Nodes
Groups:
- Intent-To-Treat: Participants received a single dose of 50 μg Lymphoseek radiolabeled with 0.5 or 1.0 mCi Tc 99m and blue dye for lymphatic mapping and surgical resection of lymph nodes.
Arm/Group | Intent-To-Treat
Number analyzed (Participants) | 136
Number analyzed (Lymph Nodes) | 215
Proportion of Lymph Nodes | 0.9767 [0.9466 to 0.9924]

2. Secondary Outcome: Reverse Concordance of Blue Dye and Lymphoseek
Description: The proportion of lymph nodes detected intraoperatively by Lymphoseek that were also detected by blue dye.
Time Frame: Surgery after injections of Lymphoseek and blue dye
Population: All enrolled patients who were injected with both Lymphoseek and blue dye, who underwent surgery and had at least one lymph node detected by Lymphoseek (at ≥ 3σ count) in vivo, and for whom the tissue type (lymphatic/non-lymphatic) and pathology status (presence/absence of tumor cells) was confirmed.
Measure: Number (95% Confidence Interval); unit: Proportion of Lymph Nodes
Units Other Than Participants: Lymph Nodes
Groups:
- Reverse Intent-To-Treat: Participants received a single dose of 50 μg Lymphoseek radiolabeled with 0.5 or 1.0 mCi Tc 99m and blue dye for lymphatic mapping and surgical resection of lymph nodes.
Arm/Group | Reverse Intent-To-Treat
Number analyzed (Participants) | 144
Number analyzed (Lymph Nodes) | 306
Proportion of Lymph Nodes | 0.6863 [0.6310 to 0.7379]

ADVERSE EVENTS:
Arm/Group | Lymphoseek
Serious Adverse Events (participants affected / at risk) | 4/179
Other Adverse Events (participants affected / at risk) | 10/179
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lymphoseek (N=179)
Myocardial Infarction (Cardiac disorders) | 1 (1) — Not related to Lymphoseek.
Nausea (Gastrointestinal disorders) | 1 (1) — Not related to Lymphoseek.
Vomiting (Gastrointestinal disorders) | 1 (1) — Not related to Lymphoseek.
Cellulitis (Infections and infestations) | 1 (1) — Not related to Lymphoseek.
Modified Radical Mastectomy (Surgical and medical procedures) | 1 (1) — Not related to Lymphoseek.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lymphoseek (N=179)
Nausea (Gastrointestinal disorders) | 10 (10) — Not related to Lymphoseek.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI shall not submit a publication to journals or professional societies without the prior written approval of the Sponsor.